CLINICAL TRIAL: NCT02575950
Title: Explorative Trial Evaluating the Efficacy and Tolerability of LEO43204 Applied in a Split-face (Left/Right) Topical Design in Adults With Moderate to Severe Acne
Brief Title: Explorative Trial Evaluating the Efficacy and Tolerability of LEO43204 in Moderate to Severe Acne
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EXP-1223
Record Dates: First submitted 2015-10-13; First posted 2015-10-15 (Estimated); Results first posted 2019-02-28 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2019-02

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- LEO43204 0,018% (Experimental): Experimental drug
  Interventions: Drug: LEO43204
- Vehicle (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LEO43204
  Arms: LEO43204 0,018%
Drug: Placebo
  Arms: Vehicle

SUMMARY:
An exploratory Phase 2, single, centre, prospective, randomized, placebo-controlled, double-blinded, split-pace (left/right) design trial to evaluate the efficacy and tolerability of LEO 43204 in adults with moderate to severe acne.

ELIGIBILITY:
Inclusion Criteria:

* Subjects should be diagnosed with acne vulgaris of the face
* Fitzpatrick skin types I-III (due to lack of safety data for the investigational product in darker skin types)
* Disease severity and total lesion count should be similar in both TAs
* Disease severity grade as moderate to severe according to the investigator's global assessment (grade 3-4)
* Age 18 to 35 years incl.
* Male or female
* Female Subjects must be of either non-childbearing potential or child-bearing potential with a confirmed negative pregnancy test

Exclusion Criteria:

* Subjects with nodulocystic acne, acne conglobata, acne fulminans, secondary acne (e.g. chlor-acne, drug-induced acne)
* Subjects with previous history of keloid formation or post-inflammatory hyperpigmentation
* Systemic retinoids within 12 month or systemic antibiotics within 1 month before Day 1
* Topical retinoids within 3 months before Day 1 or other topical treatments and/or medicated products and cosmetics that in the opinion of the investigator may influence the subjects acne vulgaris (including soaps containing antibacterial agents such as benzoyl peroxide, keratinolytic agents such as salicylic acid, skin fresheners/astringents or aftershave products) within 1 month before Day 1

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2016-06; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hala Koudsi, MD, Principal Investigator — Torrance Clinical Research Institute Inc.
Locations (1):
- Torrance Clinical Research Institute Inc., Lomita, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 19 of the participants enrolled were screening failures. The remaining 40 were enrolled sequentially into 4 cohorts. Progression from one cohort to the next was decided by the Safety Review Committee following a review of local skin responses (LSRs), safety, and tolerability after the last participant in each cohort had completed the Week 2 visit.
Groups:
- Cohort 1: Participants received once daily treatment with LEO 43204 gel 0.018% and LEO 43204 gel vehicle on either left or right cheek acne lesion areas (approx. 36 cm2 each) sequentially so that the second and third participants were not dosed until a safety evaluation of the preceding participant had been done. The first participant was dosed for 1 day, the second participant for up to 2 days, and the third participant for up to 3 days.
- Cohort 2; Cohort 4: Participants received once daily treatment with LEO 43204 gel 0.018% and LEO 43204 gel vehicle on either left or right cheek acne lesion areas of approximately 36 cm2 each for 3 days with Days 2 and 3 optional.
- Cohort 3: Participants received once daily treatment with LEO 43204 gel 0.018 and LEO 43204 gel vehicle on either left or right cheek acne lesion areas of approximately 36 cm2 each for 3 days with Days 2 and 3 optional.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Started | 3 | 6 | 6 | 25
Completed | 3 | 5 | 6 | 20
Not Completed | 0 | 1 | 0 | 5
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 1 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: All participants randomized to treatment
Arm/Group | Total
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.9 (3.8)
Age, Customized [Count of Participants; unit: Participants]
  Years: 18-20 | 18
  Years: 21-24 | 16
  Years: 25-35 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Total Lesion Count (Inflammatory and Non-inflammatory)
Description: Total lesion count (inflammatory and non-inflammatory) in acne lesion areas.
Time Frame: At Week 12 (Day 84)
Population: The analysis was based on the full analysis set (FAS). At Week 12, FAS comprised 32 subjects as 6 subjects discontinued before Week 12. The overall number of participants analyzed is irrespective of the number of participants providing data or not.
Measure: Least Squares Mean (95% Confidence Interval); unit: Lesions
Groups:
- LEO 43204 0.018%: LEO 43204 0.018% gel administered in acne lesion area either left or right cheek
- Vehicle: LEO 43204 vehicle gel administered in acne lesion area on either left or right cheek
Arm/Group | LEO 43204 0.018% | Vehicle
Number analyzed (Participants) | 38 | 38
Lesions | 23.57 [19.85 to 27.29] | 32.90 [29.18 to 36.62]
Statistical Analysis 1: Comparison: LEO 43204 0.018% vs Vehicle; Least square mean values and difference is from ANCOVA model with treatment as fixed effect and baseline total lesion count as covariate and participants as random effect. 100 simulations of monotone multiple imputation is performed. Summary statistics are found across these 100 simulations; Test type: Superiority; p < .001, ANCOVA; Mean Difference (Final Values) = -9.34, 95% CI 2-sided [-14.71 to -3.96]

2. Secondary Outcome: Inflammatory Lesion Count
Description: Count of inflammatory lesions in acne lesion areas
Time Frame: At Week 12 (Day 84)
Population: The analysis was based on the full analysis set (FAS). The FAS consisted of all participants except the first 2 participants included in Cohort 1 (according to protocol) were included in the FAS, thus the FAS comprised 38 participants. At Week 12, FAS comprised 32 participants as 6 participants discontinued before Week 12.
Measure: Mean (Standard Deviation); unit: Lesions
Groups:
- LEO 43204 0.018%: LEO 43204 0.018% gel administered in acne lesion area on either left or right cheek
Arm/Group | LEO 43204 0.018% | Vehicle
Number analyzed (Participants) | 32 | 32
Lesions | 3.81 (5.28) | 5.91 (4.55)

3. Secondary Outcome: Non-inflammatory Lesion Count
Description: Count of non-inflammatory lesions in acne lesion areas
Time Frame: At Week 12 (Day 84)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | LEO 43204 0.018% | Vehicle
Number analyzed (Participants) | 32 | 32
Lesions | 20.03 (14.25) | 25.31 (19.68)

4. Secondary Outcome: Number of Participants Stratified by Investigator's Global Assessment (IGA) of the Treatment Area
Description: The IGA score was determined according to the 5 point scale below.
  0=Clear skin with no inflammatory and non-inflammatory lesions
  1. Almost clear; rare non-inflammatory lesions with no more than one small inflammatory lesion
  2. Mild severity; greater than Grade 1; some non-inflammatory lesions with no more than a few inflammatory lesions (papules/pustules only, no nodular lesions)
  3. Moderate severity; greater than Grade 2; up to many non-inflammatory lesions and may have some inflammatory lesions, but no more than one small nodular lesions
  4. Severe; greater than Grade 3; up to many non-inflammatory and inflammatory lesions, but no more than a few nodular lesions
Time Frame: At Week 12 (Day 84)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | LEO 43204 0.018% | Vehicle
Number analyzed (Participants) | 32 | 32
Participants
  IGA score 1 | 3 | 2
  IGA score 2 | 19 | 5
  IGA score 3 | 9 | 24
  IGA score 4 | 1 | 1

5. Secondary Outcome: Composite Local Skin Response (LSR) Score at All Visits
Description: The Local Skin Responses consists of the following 6 components: erythema, flaking/scaling, crusting, swelling, vesiculation/pustulation, erosion/ulceration. Each individual LSR component is given a numeric grade of severity from 0-4. Grade 0 being no presence and Grade 4 being the highest grade of severity. The composite LSR score (0-24) is the sum of the scores graded from 0 to 4 on all six individual LSR categories.
  Please see following outcome measure descriptions on the grading scale for the individual components:
  * Erosion/ulceration: 6. Secondary outcome measure
  * Crusting: 7. Secondary outcome measure.
  * Erythema: 8. Secondary outcome measure.
  * Flaking/scaling: 9. Secondary outcome measure.
  * Swelling: 10. Secondary outcome measure.
  * Vesiculation/pustulation: 11. Secondary outcome measure.
Time Frame: At baseline (Day 1), Day 2, Day 3, Day 4, Day 8, Week 2, Week 4, Week 8 and Week 12
Population: 6 participants did not complete the trial and 7 participants had one or more missing visits during the trial.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LEO 43204 0.018% | Vehicle
Number analyzed (Participants) | 40 | 40
score on a scale
  Day 1: number analyzed (Participants) | 38 | 39
  Day 1 | 0.13 (0.81) | 0.00 (0.00)
  Day 2: number analyzed (Participants) | 38 | 39
  Day 2 | 1.34 (2.18) | 0.41 (1.50)
  Day 3: number analyzed (Participants) | 38 | 39
  Day 3 | 3.03 (2.76) | 0.90 (2.30)
  Day 4: number analyzed (Participants) | 37 | 38
  Day 4 | 4.32 (3.67) | 0.97 (2.67)
  Day 8: number analyzed (Participants) | 15 | 16
  Day 8 | 3.00 (2.62) | 0.19 (0.54)
  Week 2: number analyzed (Participants) | 35 | 36
  Week 2 | 1.17 (1.44) | 0.33 (1.24)
  Week 4: number analyzed (Participants) | 35 | 37
  Week 4 | 0.23 (0.65) | 0.05 (0.23)
  Week 8: number analyzed (Participants) | 34 | 35
  Week 8 | 0.12 (0.69) | 0.00 (0.00)
  Week 12: number analyzed (Participants) | 34 | 34
  Week 12 | 0.09 (0.38) | 0.00 (0.00)

6. Secondary Outcome: Participant's Component LSR Score: Erosion/Ulceration
Description: The Erosion/Ulceration score was determined according to the 5 point scale below.
  0=not present
  1. Lesion specific erosion
  2. Erosion extending beyond individual lesions
  3. Erosion >50%
  4. Black eschar or ulceration
Time Frame: At Day 1, Day 2, Day 3, Day 4, Day 8, Week 2, Week 4, Week 8 and Week 12
Population: 6 participants did not complete the trial and 7 participants had one or more missing visits during the trial.
Measure: Count of Participants; unit: Participants
Arm/Group | LEO 43204 0.018% | Vehicle
Number analyzed (Participants) | 40 | 40
Participants
  Day 1: number analyzed (Participants) | 38 | 39
  Day 1: Score 0 | 38 | 39
  Day 1: Score 1 | 0 | 0
  Day 1: Score 2 | 0 | 0
  Day 1: Score 3 | 0 | 0
  Day 2: number analyzed (Participants) | 38 | 39
  Day 2: Score 0 | 38 | 39
  Day 2: Score 1 | 0 | 0
  Day 2: Score 2 | 0 | 0
  Day 2: Score 3 | 0 | 0
  Day 3: number analyzed (Participants) | 38 | 39
  Day 3: Score 0 | 38 | 39
  Day 3: Score 1 | 0 | 0
  Day 3: Score 2 | 0 | 0
  Day 3: Score 3 | 0 | 0
  Day 4: number analyzed (Participants) | 37 | 38
  Day 4: Score 0 | 37 | 38
  Day 4: Score 1 | 0 | 0
  Day 4: Score 2 | 0 | 0
  Day 4: Score 3 | 0 | 0
  Day 8: number analyzed (Participants) | 15 | 16
  Day 8: Score 0 | 15 | 16
  Day 8: Score 1 | 0 | 0
  Day 8: Score 2 | 0 | 0
  Day 8: Score 3 | 0 | 0
  Week 2: number analyzed (Participants) | 35 | 36
  Week 2: Score 0 | 35 | 36
  Week 2: Score 1 | 0 | 0
  Week 2: Score 2 | 0 | 0
  Week 2: Score 3 | 0 | 0
  Week 4: number analyzed (Participants) | 35 | 37
  Week 4: Score 0 | 35 | 37
  Week 4: Score 1 | 0 | 0
  Week 4: Score 2 | 0 | 0
  Week 4: Score 3 | 0 | 0
  Week 8: number analyzed (Participants) | 34 | 35
  Week 8: Score 0 | 34 | 35
  Week 8: Score 1 | 0 | 0
  Week 8: Score 2 | 0 | 0
  Week 8: Score 3 | 0 | 0
  Week 12: number analyzed (Participants) | 34 | 34
  Week 12: Score 0 | 34 | 34
  Week 12: Score 1 | 0 | 0
  Week 12: Score 2 | 0 | 0
  Week 12: Score 3 | 0 | 0

7. Secondary Outcome: Participant's Component LSR Score: Crusting
Description: The crusting score was determined according to the 5 point scale below.
  0=not present
  1. isolated crusting
  2. Crusting<50%
  3. Crusting>50%
  4. Crusting extending outside treatment area
Time Frame: At Day 1, Day 2, Day 3, Day 4, Day 8, Week 2, Week 4, Week 8 and Week 12
Population: 6 participants did not complete the trial and 7 participants had one or more missing visits during the trial.
Measure: Count of Participants; unit: Participants
Arm/Group | LEO 43204 0.018% | Vehicle
Number analyzed (Participants) | 40 | 40
Participants
  Day 1: number analyzed (Participants) | 38 | 39
  Day 1: Score 0 | 37 | 39
  Day 1: Score 1 | 0 | 0
  Day 1: Score 2 | 1 | 0
  Day 1: Score 3 | 0 | 0
  Day 2: number analyzed (Participants) | 38 | 39
  Day 2: Score 0 | 37 | 39
  Day 2: Score 1 | 0 | 0
  Day 2: Score 2 | 0 | 0
  Day 2: Score 3 | 1 | 0
  Day 3: number analyzed (Participants) | 38 | 39
  Day 3: Score 0 | 28 | 36
  Day 3: Score 1 | 5 | 1
  Day 3: Score 2 | 5 | 1
  Day 3: Score 3 | 0 | 1
  Day 4: number analyzed (Participants) | 37 | 38
  Day 4: Score 0 | 20 | 33
  Day 4: Score 1 | 8 | 2
  Day 4: Score 2 | 6 | 2
  Day 4: Score 3 | 3 | 1
  Day 8: number analyzed (Participants) | 15 | 16
  Day 8: Score 0 | 5 | 15
  Day 8: Score 1 | 5 | 1
  Day 8: Score 2 | 5 | 0
  Day 8: Score 3 | 0 | 0
  Week 2: number analyzed (Participants) | 35 | 36
  Week 2: Score 0 | 24 | 32
  Week 2: Score 1 | 8 | 1
  Week 2: Score 2 | 3 | 2
  Week 2: Score 3 | 0 | 1
  Week 4: number analyzed (Participants) | 35 | 37
  Week 4: Score 0 | 33 | 36
  Week 4: Score 1 | 2 | 1
  Week 4: Score 2 | 0 | 0
  Week 4: Score 3 | 0 | 0
  Week 8: number analyzed (Participants) | 34 | 35
  Week 8: Score 0 | 33 | 35
  Week 8: Score 1 | 0 | 0
  Week 8: Score 2 | 1 | 0
  Week 8: Score 3 | 0 | 0
  Week 12: number analyzed (Participants) | 34 | 34
  Week 12: Score 0 | 33 | 34
  Week 12: Score 1 | 1 | 0
  Week 12: Score 2 | 0 | 0
  Week 12: Score 3 | 0 | 0

8. Secondary Outcome: Participant's Component LSR Score: Erythema
Description: The erythema score was determined according to the 5 point scale below. Erythema 0=not present
  1. slightly pink <50%
  2. Pink or light red >50%
  3. Red,restricted to treatment area
  4. Red extending outside treatment area
Time Frame: At Day 1, Day 2, Day 3, Day 4, Day 8, Week 2, Week 4, Week 8 and Week 12
Population: 6 participants did not complete the trial and 7 participants had one or more missing visits during the trial.
Measure: Count of Participants; unit: Participants
Arm/Group | LEO 43204 0.018% | Vehicle
Number analyzed (Participants) | 40 | 40
Participants
  Day 1: number analyzed (Participants) | 38 | 39
  Day 1: Score 0 | 38 | 39
  Day 1: Score 1 | 0 | 0
  Day 1: Score 2 | 0 | 0
  Day 1: Score 3 | 0 | 0
  Day 2: number analyzed (Participants) | 38 | 39
  Day 2: Score 0 | 20 | 33
  Day 2: Score 1 | 8 | 3
  Day 2: Score 2 | 6 | 2
  Day 2: Score 3 | 4 | 1
  Day 3: number analyzed (Participants) | 38 | 39
  Day 3: Score 0 | 9 | 31
  Day 3: Score 1 | 11 | 2
  Day 3: Score 2 | 13 | 3
  Day 3: Score 3 | 5 | 3
  Day 4: number analyzed (Participants) | 37 | 38
  Day 4: Score 0 | 10 | 33
  Day 4: Score 1 | 8 | 1
  Day 4: Score 2 | 9 | 1
  Day 4: Score 3 | 10 | 3
  Day 8: number analyzed (Participants) | 15 | 16
  Day 8: Score 0 | 9 | 16
  Day 8: Score 1 | 4 | 0
  Day 8: Score 2 | 1 | 0
  Day 8: Score 3 | 1 | 0
  Week 2: number analyzed (Participants) | 35 | 36
  Week 2: Score 0 | 31 | 35
  Week 2: Score 1 | 3 | 1
  Week 2: Score 2 | 1 | 0
  Week 2: Score 3 | 0 | 0
  Week 4: number analyzed (Participants) | 35 | 37
  Week 4: Score 0 | 34 | 37
  Week 4: Score 1 | 1 | 0
  Week 4: Score 2 | 0 | 0
  Week 4: Score 3 | 0 | 0
  Week 8: number analyzed (Participants) | 34 | 35
  Week 8: Score 0 | 34 | 35
  Week 8: Score 1 | 0 | 0
  Week 8: Score 2 | 0 | 0
  Week 8: Score 3 | 0 | 0
  Week 12: number analyzed (Participants) | 34 | 34
  Week 12: Score 0 | 34 | 34
  Week 12: Score 1 | 0 | 0
  Week 12: Score 2 | 0 | 0
  Week 12: Score 3 | 0 | 0

9. Secondary Outcome: Participant's Component LSR Score: Flaking/Scaling
Description: The flaking/scaling score was determined according to the 5 point scale below. 0=not present
  1. Isolated scale, specific to lesion
  2. Scale<50%
  3. Scale>50%
  4. Scaling extending outside treatment area
Time Frame: At Day 1, Day 2, Day 3, Day 4, Day 8, Week 2, Week 4, Week 8 and Week 12
Population: 6 participants did not complete the trial and 7 participants had one or more missing visits during the trial.
Measure: Count of Participants; unit: Participants
Arm/Group | LEO 43204 0.018% | Vehicle
Number analyzed (Participants) | 40 | 40
Participants
  Day 1: number analyzed (Participants) | 38 | 39
  Day 1: Score 0 | 37 | 39
  Day 1: Score 1 | 0 | 0
  Day 1: Score 2 | 0 | 0
  Day 1: Score 3 | 1 | 0
  Day 2: number analyzed (Participants) | 38 | 39
  Day 2: Score 0 | 37 | 39
  Day 2: Score 1 | 1 | 0
  Day 2: Score 2 | 0 | 0
  Day 2: Score 3 | 0 | 0
  Day 3: number analyzed (Participants) | 38 | 39
  Day 3: Score 0 | 25 | 36
  Day 3: Score 1 | 10 | 2
  Day 3: Score 2 | 3 | 1
  Day 3: Score 3 | 0 | 0
  Day 4: number analyzed (Participants) | 37 | 38
  Day 4: Score 0 | 15 | 32
  Day 4: Score 1 | 11 | 3
  Day 4: Score 2 | 7 | 2
  Day 4: Score 3 | 4 | 1
  Day 8: number analyzed (Participants) | 15 | 16
  Day 8: Score 0 | 3 | 14
  Day 8: Score 1 | 8 | 2
  Day 8: Score 2 | 4 | 0
  Day 8: Score 3 | 0 | 0
  Week 2: number analyzed (Participants) | 35 | 36
  Week 2: Score 0 | 19 | 35
  Week 2: Score 1 | 11 | 0
  Week 2: Score 2 | 5 | 0
  Week 2: Score 3 | 0 | 1
  Week 4: number analyzed (Participants) | 35 | 37
  Week 4: Score 0 | 30 | 36
  Week 4: Score 1 | 5 | 1
  Week 4: Score 2 | 0 | 0
  Week 4: Score 3 | 0 | 0
  Week 8: number analyzed (Participants) | 34 | 35
  Week 8: Score 0 | 33 | 35
  Week 8: Score 1 | 0 | 0
  Week 8: Score 2 | 1 | 0
  Week 8: Score 3 | 0 | 0
  Week 12: number analyzed (Participants) | 34 | 34
  Week 12: Score 0 | 33 | 34
  Week 12: Score 1 | 1 | 0
  Week 12: Score 2 | 0 | 0
  Week 12: Score 3 | 0 | 0

10. Secondary Outcome: Participant's Component LSR Score: Swelling
Description: The swelling score was determined according to the 5 point scale below. 0=Not present
  1. Slight, lesion specific oedema
  2. Palpable oedema extending beyond individual lesions
  3. Confluent and/or visible oedema
  4. Marked swelling extending outside treatment area
Time Frame: At Day 1, Day 2, Day 3, Day 4, Day 8, Week 2, Week 4, Week 8 and Week 12
Population: 6 participants did not complete the trial and 7 participants had one or more missing visits during the trial.
Measure: Count of Participants; unit: Participants
Arm/Group | LEO 43204 0.018% | Vehicle
Number analyzed (Participants) | 40 | 40
Participants
  Day 1: number analyzed (Participants) | 38 | 39
  Day 1: Score 0 | 38 | 39
  Day 1: Score 1 | 0 | 0
  Day 1: Score 2 | 0 | 0
  Day 1: Score 3 | 0 | 0
  Day 2: number analyzed (Participants) | 38 | 39
  Day 2: Score 0 | 32 | 38
  Day 2: Score 1 | 2 | 0
  Day 2: Score 2 | 3 | 1
  Day 2: Score 3 | 1 | 0
  Day 3: number analyzed (Participants) | 38 | 39
  Day 3: Score 0 | 25 | 37
  Day 3: Score 1 | 7 | 1
  Day 3: Score 2 | 6 | 1
  Day 3: Score 3 | 0 | 0
  Day 4: number analyzed (Participants) | 37 | 38
  Day 4: Score 0 | 27 | 37
  Day 4: Score 1 | 8 | 1
  Day 4: Score 2 | 2 | 0
  Day 4: Score 3 | 0 | 0
  Day 8: number analyzed (Participants) | 15 | 16
  Day 8: Score 0 | 14 | 16
  Day 8: Score 1 | 1 | 0
  Day 8: Score 2 | 0 | 0
  Day 8: Score 3 | 0 | 0
  Week 2: number analyzed (Participants) | 35 | 36
  Week 2: Score 0 | 35 | 36
  Week 2: Score 1 | 0 | 0
  Week 2: Score 2 | 0 | 0
  Week 2: Score 3 | 0 | 0
  Week 4: number analyzed (Participants) | 35 | 37
  Week 4: Score 0 | 35 | 37
  Week 4: Score 1 | 0 | 0
  Week 4: Score 2 | 0 | 0
  Week 4: Score 3 | 0 | 0
  Week 8: number analyzed (Participants) | 34 | 35
  Week 8: Score 0 | 34 | 35
  Week 8: Score 1 | 0 | 0
  Week 8: Score 2 | 0 | 0
  Week 8: Score 3 | 0 | 0
  Week 12: number analyzed (Participants) | 34 | 34
  Week 12: Score 0 | 34 | 34
  Week 12: Score 1 | 0 | 0
  Week 12: Score 2 | 0 | 0
  Week 12: Score 3 | 0 | 0

11. Secondary Outcome: Participant's Component LSR Score: Vesiculation/Pustulation
Description: The vesiculation/postulation score was determined according to the 5 point scale below.
  0=not present
  1. vesicles only
  2. Transudate or pustulates with or without vesicles <50%
  3. Transudate or pustulates, with or without vesicles >50%
  4. Transudate or pustulates, with or without vesicles extending outside treatment area
  4=Marked swelling extending outside treatment area
Time Frame: At Day 1, Day 2, Day 3, Day 4, Day 8, Week 2, Week 4, Week 8 and Week 12
Population: 6 participants did not complete the trial and 7 participants had one or more missing visits during the trial.
Measure: Count of Participants; unit: Participants
Arm/Group | LEO 43204 0.018% | Vehicle
Number analyzed (Participants) | 40 | 40
Participants
  Day 1: number analyzed (Participants) | 38 | 39
  Day 1: Score 0 | 38 | 39
  Day 1: Score 1 | 0 | 0
  Day 1: Score 2 | 0 | 0
  Day 1: Score 3 | 0 | 0
  Day 2: number analyzed (Participants) | 38 | 38
  Day 2: Score 0 | 36 | 38
  Day 2: Score 1 | 1 | 0
  Day 2: Score 2 | 0 | 0
  Day 2: Score 3 | 1 | 0
  Day 3: number analyzed (Participants) | 38 | 39
  Day 3: Score 0 | 30 | 37
  Day 3: Score 1 | 4 | 0
  Day 3: Score 2 | 3 | 1
  Day 3: Score 3 | 1 | 1
  Day 4: number analyzed (Participants) | 37 | 38
  Day 4: Score 0 | 24 | 36
  Day 4: Score 1 | 4 | 0
  Day 4: Score 2 | 5 | 1
  Day 4: Score 3 | 4 | 1
  Day 8: number analyzed (Participants) | 15 | 16
  Day 8: Score 0 | 13 | 16
  Day 8: Score 1 | 1 | 0
  Day 8: Score 2 | 0 | 0
  Day 8: Score 3 | 1 | 0
  Week 2: number analyzed (Participants) | 35 | 36
  Week 2: Score 0 | 34 | 36
  Week 2: Score 1 | 1 | 0
  Week 2: Score 2 | 0 | 0
  Week 2: Score 3 | 0 | 0
  Week 4: number analyzed (Participants) | 35 | 37
  Week 4: Score 0 | 35 | 37
  Week 4: Score 1 | 0 | 0
  Week 4: Score 2 | 0 | 0
  Week 4: Score 3 | 0 | 0
  Week 8: number analyzed (Participants) | 34 | 35
  Week 8: Score 0 | 34 | 35
  Week 8: Score 1 | 0 | 0
  Week 8: Score 2 | 0 | 0
  Week 8: Score 3 | 0 | 0
  Week 12: number analyzed (Participants) | 34 | 34
  Week 12: Score 0 | 33 | 34
  Week 12: Score 1 | 1 | 0
  Week 12: Score 2 | 0 | 0
  Week 12: Score 3 | 0 | 0

12. Secondary Outcome: Number of Participants With Occurrence of Unacceptable LSR Scores or Unacceptable Safety and Tolerability Events at All Visits
Description: Unacceptable LSRs, safety and tolerability in an individual participant were defined as:
  1. Clinically relevant signs or symptoms that in the opinion of the investigator were deemed unacceptable.
  2. Occurrence of LSRs as specified below:
  One of the following
  * Grade 4 crusting
  * Grade 4 erosion/ulceration
  * Grade 4 vesiculation/pustulation extending significantly outside treatment areas
  Two of the following
  * Grade 4 erythema
  * Grade 3 crusting
  * Grade 4 swelling extending significantly outside treatment areas
  * Grade 3 erosion/ulceration
  * Grade 3 vesiculation/pustulation
Time Frame: At Day 1, Day 2, Day 3, Day 4, Day 8, Week 2, Week 4, Week 8 and Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | LEO 43204 0.018% | Vehicle
Number analyzed (Participants) | 40 | 40
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: From baseline (Day 1) to post treatment follow-up (end of treatment to Week 12)
Groups:
- Non-cutaneous: Non-cutaneous adverse events
- LEO 43204 0.018%: LEO 43204 0.018% gel administered to an acne lesion on either left or right cheek
- Vehicle: LEO 43204 vehicle gel administered to an acne lesion on either left or right cheek
Arm/Group | Non-cutaneous | LEO 43204 0.018% | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 2/40 | 18/40 | 1/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-cutaneous (N=40) | LEO 43204 0.018% (N=40) | Vehicle (N=40)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Application site pruritus (General disorders) | 0 (0) | 2 (2) | 0 (0)
Application site pain (General disorders) | 0 (0) | 18 (18) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
LEO acknowledges the investigators right to publish the entire results of the study, irrespective of outcome. LEO retains the right to have any publication submitted to LEO for review. Investigators must undertake not to submit any part of their individual data for publication without the prior consent of LEO.

DOCUMENTS (2):
  • Study Protocol (2016-09-15): https://cdn.clinicaltrials.gov/large-docs/50/NCT02575950/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-19): https://cdn.clinicaltrials.gov/large-docs/50/NCT02575950/SAP_001.pdf